CLINICAL TRIAL: NCT02301507
Title: Evaluation of Texting Intervention to Improve Adherence to Antiretroviral Therapy (ART) in Young Women Infected With Human Immunodeficiency Virus (HIV)
Brief Title: Study of Cell Phone SMS to Improve Adherence to ART in HIV Positive Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Tanvir K. Bell, MD, Associate Professor of Medicine, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-14-0692
Record Dates: First submitted 2014-11-18; First posted 2014-11-26 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SMS (texting) Arm (Experimental): texts received
  Interventions: Behavioral: cell phone SMS text messaging

INTERVENTIONS:
Behavioral: cell phone SMS text messaging — This study will utilize mobile texting services to send text messages to enrolled subjects on a weekly basis. The text would convey messages that promote better awareness and knowledge on HIV and its treatment, reminders for medication adherence and clinic appointments. The text content would also be customized based on individual subject requirements. English will be used in texting. We would also assess the subjects for traditional demographic items (e.g., age, marital status, education, number/age of other children, employment, and religion), and potential environmental barriers (e.g., transportation and childcare).

SUMMARY:
There has been increasing use of technology in delivery of healthcare and increasing use of cellular phone and text messaging services to help with various healthcare related issues including but not limited to medication adherence and clinic attendance. Mobile phones technology has been used for healthcare delivery and prevention strategies such as smoking cessation. In the present era, cell phones have become part of daily life for most people even among those in lower economic groups. There have also been several studies looking at cell phone text messaging services to improve adherence to ART among HIV infected subjects but no studies have so far been done in HIV infected young women to help retention and adherence to care. The overall goal of this study is to evaluation of the impact of texting intervention to improve adherence to care and treatment in HIV infected young women.

Study Hypothesis:

Text message intervention will improve adherence to ART in HIV infected young women.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected women who have been newly diagnosed within the past 1 year or who are just entering into care at Thomas Street Health Center.
2. Subjects must be 18 years or older.
3. Subjects must have cell phones with texting capability.
4. Ability to speak, read, or understand English or Spanish.
5. Must be willing and able to respond to text messages.

Exclusion Criteria:

1. Women who are unable to speak, read, or understand English or Spanish

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Improve adherence to care and treatment in HIV infected young women. The outcome measure will be assessed by capturing kept medical appointments. | 6 months

SECONDARY OUTCOMES:
assess improvements in stigma and depression in HIV infected women. The outcome measure will be assessed by questionaires. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Street Health Center, Houston, Texas, United States